CLINICAL TRIAL: NCT02541799
Title: Comprehension of Research Informed Consent When Applied Through a Telemedicine Medium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Mohr, Nicholas M, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201504742
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Informed Consent
Keywords: informed consent; telemedicine; research methods
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine (Experimental): Participants allocated to this arm will be approached the using a telemedicine medium to discuss study participation. The consent form will be administered while the investigator is on a telemedicine link.
  Interventions: Procedure: Audio-visual telemedicine
- Standard Care (Active Comparator): Participants allocated to this arm will be approached in standard fashion where the investigator approaches the patient face to face. The consent form will be administered while the investigator is in the participant's room.
  Interventions: Procedure: Standard care

INTERVENTIONS:
Procedure: Audio-visual telemedicine — Participants in an emergency department will have their care delivered using telemedicine, then they will be approached for a study by a study investigator using the same telemedicine link
  Arms: Telemedicine
Procedure: Standard care — Participants in an emergency department will have their care delivered in person, then they will be approached by a study investigator face-to-face.
  Arms: Standard Care

SUMMARY:
The investigators hypothesis is that patient comprehension of telemedicine-enabled research informed consent is not inferior to standard face-to-face research informed consent.

The procotol will involve a prospective, randomized control trial to test the effectiveness of a telemedicine medium in obtaining research informed consent. Within a single emergency department, the investigators will conduct a simple, low risk randomized trial (single does of oral chlorhexideine to prevent hospital acquired pneumonia among adult patients with expected hospital admission). Prior to being approached for informed consent, potential participants will be randomized in a 1:1 allocation ratio to standard face-to-face consent vs. consent provided by audio-visual telemedicine. After standard clinical care, potential participants will be approached according to their allocation. Comprehension of research informed consent will be the primary outcome, and will be measured using the modified Quality of Informed Consent (QuIC) instrument.

ELIGIBILITY:
Inclusion Criteria:

* any adult patient presenting to the emergency department, and expected to be admitted to the hospital.

Exclusion Criteria:

* prisoners
* pregnant patients
* non-English speaking patients
* unable to provide informed consent based on mental status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Comprehension of research informed consent | Immediately
  Comprehension of research informed consent will be assessed within 30 minutes of approaching participants for study inclusion. The QuIC will be used to assess comprehension of the elements of research informed consent.

SECONDARY OUTCOMES:
Consent rate | Immediately
  Rate of consenting for a low-risk clinical trial in the emergency department, depending on how research participation was solicited.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States